CLINICAL TRIAL: NCT05376410
Title: Relationship Between Maternal Soluble Trigger Receptor Expressed on Myeloid Cells-1 (sTREM-1) and Placenta Accreta Spectrum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hasan Energin, asistan professor, Necmettin Erbakan University
Other Study IDs: NecmettinErbakanUniversity
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Placenta Accreta, Third Trimester
Keywords: Placenta Accreta, sTREM-1
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We planed to evaluate soluble the triggering receptors expressed on myeloid cell-1 (s TREM-1) levels in serum of pregnant women diagnosed with placenta accreta spectrum and compare it with healthy pregnant women's s TREM-1 serum levels.

DETAILED DESCRIPTION:
Placenta accreta, which was a rare diagnosis before, is now one of the most important causes of postpartum hemorrhage and hysterectomy. Trigger receptor expressed on myeloid cells (TREM), interacts with Toll-like receptors (TLRs) that play an important role in the immune response (TLRs are found in many immune system cells, such as natural killer cells, macrophages, lymphocytes), and TLR-induced signaling modulates the incoming immune response by amplifying or suppressing it. One of the most appealing features of the TREM family is the release of soluble receptors. Soluble TREM-1 (sTREM-1) is a 17-kDa fragment; which is hypothesized to be pro- duced by alternative splicing of the Trem 1 gene or by proteolytic cleavage by metalloproteinases (MMPs).

Although major risk factors of placenta accreta are previous cesarian deliverers and placenta previa It can be seen in nulliparous women without any low lying placenta. The pathophysiology of the disease is still unknown. Some authors hypothesized that immune system play role in its pathophysiology.

We planed to evaluate soluble the triggering receptors expressed on myeloid cell-1 (s TREM-1) levels in serum of pregnant women diagnosed with placenta accreta spectrum and compare it with healthy pregnant women's s TREM-1 serum levels.

The study is planned as a case control study. 30 pregnant women diagnosed with placenta accreta and 60 healthy pregnant women will be included in the study. The study is planned to last 9 months in total. TREM-1 will be studied from the blood taken routinely from the participants during their follow-up in the outpatient clinic or service.

Inclusion criteria for the study were determined as being in the 3rd trimester, not having any additional disease, not in labor, not having multiple pregnancy.

Exclusion criteria: Not being at the specified gestational week, having multiple pregnancy, having any additional disease, having an infection, being in labor.

After the diagnosis of placenta accreta , a 5 cm3 of venous blood samples of the patients will be collected from their antecubital veins after 12h of fasting in 24h. Serum samples will be isolated by centrifugation at 3000rpm for min. The samples will be maintained at 80C before performing assays. Serum triggering receptor expressed on myeloid cells 1 concentrations will be measured using a commercially available enzyme- linked immunosorbent assay (ELISA) kit.

ELIGIBILITY:
Inclusion Criteria: placenta accreta spectrum diagnosis. 3rd trimester pregnancy, not having any additional disease, not in labor, not having multiple pregnancy.

Exclusion Criteria:having multiple pregnancy, having any additional disease (preeclampsia, gestational diabetes mellitus, etc) , having an infection, being in labor.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant.
Study Population: 3rd trimester pregnancies diagnosed with placenta accreta spectrum.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
sTREM-1 levels | after 12 hours fasting
  sTREM-1 levels in maternal serum

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Meram Medicine Faculty, Konya, Turkey (Türkiye)